CLINICAL TRIAL: NCT01689038
Title: Brain Imaging Study of F17464
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: F17464 PO 1 02
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — dopamine D3 receptor antagonist F17464

ARMS (1):
- Tested product (Experimental)
  Interventions: Drug: F17464

INTERVENTIONS:
Drug: F17464 — Single dose

SUMMARY:
Assess the binding rate of F17464 to cerebral receptors in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers

Exclusion Criteria:

* Presence or positive history of severe medical illness or psychiatric conditions

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Binding rate to cerebral receptors | up to 29 hours
  by brain imaging

CONTACTS AND LOCATIONS:
Locations (1):
- New York, New York, United States